CLINICAL TRIAL: NCT06593093
Title: A Bundled Intervention to End Opioid Overdose by Increasing Treatment Uptake Post Emergency Department Discharge
Brief Title: A Bundled Intervention
Acronym: B-CARE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Li Li, Full Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300013272; R61DA062351 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder; Opioid Overdose
Keywords: Emergency department; post discharge; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Emergencies | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- phase 1 (Experimental): After completing screening questions and obtaining consent, eligible participants will complete their baseline procedures and measures. All participants will then start the experimental, i.e., bundled intervention, the first week after their ED discharge, including peer support service and buprenorphine treatment with addiction physicians using telehealth. Each participant will be in the study for 3 months. During the study period, participants will be sent survey links to their cell phones and/or emails to complete self-report questionnaires via the Research Electronic Data Capture (REDCap) at 1-month and 3-month for follow-up assessments. Peers will remind the participants to complete the survey.
  Interventions: Other: a bundled intervention
- phase 2- experimental (Experimental): Participants will be enrolled the same way as in phase 1. After their enrollment, participants will be randomized to either the experimental (bundled intervention) group or the control (usual care group). Bundled intervention will have the same components as in the phase 1, including peer support, buprenorphine treatment, and telehealth up to 3 months after ED/hospital discharge, and linkage to definitive addiction treatment programs. Participants will be sent survey links to their cell phones and emails to complete self-report questionnaires via REDCap at 1- and 3-month for follow-up assessments. Participants will be reminded via text messages and/or emails to complete the survey twice per day 5 days prior to their follow-up assessments.
  Interventions: Other: a bundled intervention
- phase 2- control (Placebo Comparator): Participants who are randomized to the control group will receive the usual care that has been established in the ED at UAB hospital. The current usual care at the UAB ED includes a thorough assessment, buprenorphine initiation as appropriate, peer referral, and a written list of buprenorphine clinics. Participants will also receive information about community-based substance use treatment programs. However, these services are at the participant's own discretion to navigate and attend after ED discharge. Participants will be sent survey links to their cell phones and emails to complete self-report questionnaires via REDCap at 1- and 3-month for follow-up assessments. Participants will be reminded via text messages and/or emails to complete the survey twice per day 5 days prior to their follow-up assessments.
  Interventions: Other: control group

INTERVENTIONS:
Other: a bundled intervention — a bundled intervention, including peer support, buprenorphine (ranging from 4mg-24mg, oral, daily), telehealth, and community-based addiction programs.
  Arms: phase 1; phase 2- experimental
Other: control group — participants will not be intervened with this bundled treatment, but continue the usual care that has been established at UAB ED.
  Arms: phase 2- control

SUMMARY:
Opioid overdose deaths have reached historically high records in the United States and are particularly concentrated among patients after emergency department (ED) discharge. Evidence-based treatment modules to reduce repeat opioid overdose and mortality are lacking in this patient population. A bundled intervention is proposed, including telehealth, peer support specialist, buprenorphine, and linkage for definitive care, that is designed to increase treatment uptake in this patient population post-ED discharge, reduce repeat opioid overdoses, and end overdose deaths.

DETAILED DESCRIPTION:
This study is supported by the HEAL Initiative (https://heal.nih.gov). Opioid overdose deaths have reached historically high records in the U.S. and are particularly concentrated among patients after emergency department (ED) discharge. Medications for opioid use disorder (MOUDs), including buprenorphine, are the most effective treatments for opioid use disorder (OUD) as MOUD reduce opioid-related overdoses and deaths. Despite this, less than 30% patients with OUD are treated with MOUDs. Furthermore, adequate treatment with MOUD can be more difficult in certain patient population, i.e., patients with nonfatal opioid overdoses after ED discharge. This patient population also accounts for substantial health care utilization, frequent ED visits, and the largest at-risk group for repeat overdoses and even deaths. Many barriers, including patients' stigma on MOUDs, lack of appropriate monitoring and support, difficulty in navigating community-based treatment programs and being connected with buprenorphine clinics for continuity of care, have been identified as contributors to poor treatment uptake post-ED discharge. These barriers present a pressing need to develop novel treatment modules. Peer support models and telehealth have been successful in improving service provision and increasing treatment uptake in substance use disorders. However, it remains untested if a bundled intervention of telehealth, peers, buprenorphine, and linkage to definitive addiction programs can increase treatment uptake in this particular population. Thus, the purpose of this proposal is to test this bundled intervention specifically focusing on patients with OUD and nonfatal opioid overdoses post-ED discharge. In the R61 phase, 30 patients with OUD and opioid overdoses in the past 12 months will be enrolled from the University of Alabama at Birmingham Hospital when participants are discharged from the ED. Following ED discharge, peers will contact patients daily in Week 1 post-ED discharge, twice in Week 2, and weekly thereafter for 12 weeks using telehealth. Physicians will continue prescribing buprenorphine. Peers will also motivate and assist participants to engage in community-based treatment programs for continuity of care after intervention is completed. Primary outcomes will be the feasibility and acceptability of this bundled intervention. In the R33 phase, participants will be enrolled and randomized to either the intervention group (N=80) or the usual care group (UC, N=80). Patients will be enrolled from the same ED and same eligibility criteria as in the R61 phase will be applied. In the intervention group, peers and physicians will provide the same intervention to patients as in the R61 phase. Patients in the UC group will receive the usual care that has been established at the ED, including ED-initiated buprenorphine, and a list of community-based substance treatment programs and buprenorphine clinics at ED discharge. However, no further intervention will be provided in the UC group. Primary outcomes will be increased treatment uptake and retention after ED discharge, and reduced opioid overdoses and ED revisits, compared to the UC group. If successful, this project will lay the groundwork for a multi-site trial to validate the treatment and to identify actual implementation and sustainability barriers and best practices.

ELIGIBILITY:
Inclusion Criteria:

1. discharged from the ED and inpatient settings at the UAB hospital
2. 19 years or older (the age of majority in Alabama);
3. diagnosis of OUD and experiencing opioid overdose in the last 12 months;
4. prescribed buprenorphine in the ED and willing to continue buprenorphine post-ED discharge;
5. English speaking;
6. not actively psychotic and suicidal, or cognitively impaired.
7. Patients who are admitted to the hospital from the ED will be eligible for enrollment.

Exclusion Criteria:

1. living in a restricted environment (e.g., prison or jail facility, etc.);
2. currently enrolled in other clinical studies;
3. anticipated to take other prescribed opioids except buprenorphine for a medical condition longer than three months;
4. known allergic reaction to buprenorphine;
5. critically ill or injured;
6. females with pregnancy (they are anticipated to request a higher level of care).
7. living outside of Alabama

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
participant retention rate | 1 month and 3 months post ED discharge
  measure the total number of participants who complete 1- month and 3-month treatment in the study
buprenorphine adherent rate | 1 month and 3 months post ED discharge
  checking prescription rate and patients' report of their taking medication rate
linkage rate to addiction treatment programs | 1 month and 3 months post ED discharge
  patients' self report and reports from addiction treatment programs

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD;PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share our data using: Conference presentations; Publications; A press release; sharing with other emergency departments across the U.S; prepare and submit subsequent grants to communicate the results of this study and to facilitate broad implementation activities; the results of this study also will be posted publicly via ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF